CLINICAL TRIAL: NCT05058820
Title: Effects of Post Facilitation Stretch Versus Active Isolated Stretching Along With Deep Friction Massage in Wallet Sciatica.
Brief Title: Post Facilitation Stretch Versus Active Isolated Stretching Along With Deep Friction Massage in Wallet Sciatica.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0971 Samira Sabir
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Wallet Sciatica
Keywords: Active Isolated stretching; Deep friction massage; Post Facilitation stretching; Piriformis syndrome
MeSH Terms: conditions — Hip socket neuropathy; Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Facilitation stretch (Experimental): Hot pack, TENS, Post Facilitation stretch, Deep friction massage
  Interventions: Other: Post Facilitation stretch
- Active Isolated Stretching (Active Comparator): Hot pack, TENS, Active Isolated Stretching, Deep friction massage
  Interventions: Other: Active Isolated Stretching

INTERVENTIONS:
Other: Post Facilitation stretch — Hot pack 10 mins/ 1set/ (3 days/ week), TENS 10 mins/ 1 set/ (3 days/ week), Post facilitation stretch 15 secs isometric hold/ 15 secs stretch/ 30 secs relax/ 5 reps/ 1 set/ (3 days/ week), Deep friction massage 5 minutes/ (3 days/ week). A total of 6 weeks (18 sessions, 3 days/ week) were given each consisting of 30 mins.
  Arms: Post Facilitation stretch
Other: Active Isolated Stretching — Hot pack 10 mins/ 1set/ (3 days/ week), TENS 10 mins/ 1 set/ (3 days/ week), Active Isolated Stretching 2 secs hold/ 10 reps/ 1 set/ (3 days/ week), Deep friction massage 5 minutes/ (3 days/ week). A total of 6 weeks (18 sessions, 3 days/ week) were given each consisting of 30 mins.
  Arms: Active Isolated Stretching

SUMMARY:
To compare the effects of post facilitation stretch and active isolated stretch along with deep friction massage on pain pressure threshold of trigger points, disability, muscle length, and hip joint range of motion in wallet sciatica.

DETAILED DESCRIPTION:
Literature shows the effectiveness of both techniques post facilitation stretch and active isolated stretch but didn't report any comparison. In this study, investigator diagnosed the patients with wallet sciatica who came with the complaint of low back pain. Both techniques were compared to determine the effectiveness in patients with wallet sciatica having trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Pain (Grade greater than 3)
* Chronic pain (greater than 3 months) buttock pain.
* Patients with piriformis tightness less than 40 degrees.
* Patients with active trigger points of the piriformis.

Exclusion Criteria:

* Patient with tumor
* Patients with cognitive problems.
* Recent or history of hip trauma or injury.
* Recent abdominal surgery.
* Any other orthopedic or neurological condition of hip and lumbar spine

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold | 18 days
  Changes from baseline, Pain pressure threshold was measured through Algometer.
Disability | 18 days
  Changes from baseline, Disability was measured through lower extremity functional scale. It consists of 20 questions. Minimum score is 0 and Maximum 80. minimum score shows greater disability and maximum indicate decreased disability.
Piriformis Muscle Length | 18 days
  Changes from baseline, Piriformis Muscle Length was measured through Goniometer by performing stretch test. Less than 40 degree internal rotation at hip indicates piriformis tightness.
Hip joint range of motion | 18 days
  Changes from baseline, Hip joint range of motion was measured through Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Momena Shahzad, MS-OMPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Ali Ahmad Physio Care, F-7/2, Islamabad, Fedral
  - Railway General Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No